CLINICAL TRIAL: NCT00168597
Title: Should Infants Receive High-dose Vitamin A Supplementation With BCG Vaccine at Birth in Developing Countries?
Brief Title: Vitamin A With BCG Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Leiden University Medical Center (Other); Medical Research Council Unit, The Gambia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICA-CT-2001-10095-VITA; ICA-CT-2001-10095
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Mortality; Morbidity
Keywords: Vitamin A; BCG; Infant mortality; Morbidity; Low-income country
MeSH Terms: conditions — Infant Death | interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
Two studies from Asia have suggested a beneficial effect of vitamin A supplementation given at birth. Hypotheses: Vitamin A supplementation administered at birth together with BCG vaccination is associated with a 30% reduction in infant mortality and morbidity during the first year of life in normal birth weight children in an African setting.

DETAILED DESCRIPTION:
Vitamin A deficiency is common in low-income countries. Vitamin A supplementation to children above 6 months of age reduces all-cause mortality with 23 % to 30 %. Studies on vitamin A supplementation in infants younger than 6 months of age have reported inconsistent effects on mortality. Studies providing supplementation between 1 and 5 months of age have found no effect or even a negative effect. However, the only two studies of supplementation at birth, both conducted in Asia, showed substantial significant reductions in infant all-cause mortality.

The beneficial effect of neonatal vitamin A supplementation may be a result of correcting the congenital vitamin A deficiency resulting from maternal vitamin A deficiency. On the other hand, it has been speculated that the beneficial effect of vitamin A supplementation given at birth may in part be explained by a synergistic effect of vitamin A supplementation and BCG vaccination given at the time of birth.

The protective effect on mortality of vitamin A supplementation given at birth needs to be confirmed in an African population. Furthermore, none of the two previous studies have reported data on vaccination status of the included infants.

In this study, the effect on mortality and morbidity of given vitamin A supplementation simultaneously with BCG vaccination at birth to normal birth weight infants will be investigated in an African population. Furthermore, the effects of vitamin A supplementation will be evaluated with respect to effect on growth, the response to BCG vaccination, infant vitamin A status and infant cytokine profile. Furthermore the effect on specific diseases such as malaria, measles and rotavirus infections. The mechanisms behind the effects of vitamin A will be evaluated.

We will include 4,800 normal birth weight infants (> 2500 g) infants randomized to 50,000 IU of vitamin A or placebo given simultaneously with BCG vaccine. The study take place in Guinea-Bissau, West Africa. The study area consists of five districts in the capital of Guinea-Bissau. The Bandim Health Project has been working in the study area for almost 25 years, and a demographic surveillance system has been established and functioned for many years.

ELIGIBILITY:
Inclusion Criteria: Belonging to the study area

Exclusion Criteria:Overt illness, signs of vitamin A deficiency, previous BCG vaccination

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4800
Dates: Start 2002-08; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mortality
Hospitalisations

SECONDARY OUTCOMES:
Adverse effects
Tuberculin reaction
BCG scarring
Growth
Vitamin A status
Cytokine responses
Malaria
Measles
Rotavirus
All primary and secondary outcomes will be analysed for interactions between vitamin A and sex and last vaccine received

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Aage S, Kiraly N, Da Costa K, Byberg S, Bjerregaard-Andersen M, Fisker AB, Aaby P, Benn CS. Neonatal vitamin A supplementation associated with increased atopy in girls. Allergy. 2015 Aug;70(8):985-94. doi: 10.1111/all.12641. Epub 2015 May 18. PMID 25939706
- [Derived] Benn CS, Martins CL, Fisker AB, Diness BR, Garly ML, Balde I, Rodrigues A, Whittle H, Aaby P. Interaction between neonatal vitamin A supplementation and timing of measles vaccination: a retrospective analysis of three randomized trials from Guinea-Bissau. Vaccine. 2014 Sep 22;32(42):5468-74. doi: 10.1016/j.vaccine.2014.07.090. Epub 2014 Aug 13. PMID 25131735
- [Derived] Fisker AB, Aaby P, Rodrigues A, Frydenberg M, Bibby BM, Benn CS. Vitamin A supplementation at birth might prime the response to subsequent vitamin A supplements in girls. Three year follow-up of a randomized trial. PLoS One. 2011;6(8):e23265. doi: 10.1371/journal.pone.0023265. Epub 2011 Aug 11. PMID 21853099
- [Derived] Diness BR, Christoffersen D, Pedersen UB, Rodrigues A, Fischer TK, Andersen A, Whittle H, Yazdanbakhsh M, Aaby P, Benn CS. The effect of high-dose vitamin A supplementation given with bacille Calmette-Guerin vaccine at birth on infant rotavirus infection and diarrhea: a randomized prospective study from Guinea-Bissau. J Infect Dis. 2010 Sep 1;202 Suppl:S243-51. doi: 10.1086/653569. PMID 20684711
- [Derived] Benn CS, Diness BR, Roth A, Nante E, Fisker AB, Lisse IM, Yazdanbakhsh M, Whittle H, Rodrigues A, Aaby P. Effect of 50,000 IU vitamin A given with BCG vaccine on mortality in infants in Guinea-Bissau: randomised placebo controlled trial. BMJ. 2008 Jun 21;336(7658):1416-20. doi: 10.1136/bmj.39542.509444.AE. Epub 2008 Jun 16. PMID 18558641
- [Derived] Diness BR, Fisker AB, Roth A, Yazdanbakhsh M, Sartono E, Whittle H, Nante JE, Lisse IM, Ravn H, Rodrigues A, Aaby P, Benn CS. Effect of high-dose vitamin A supplementation on the immune response to Bacille Calmette-Guerin vaccine. Am J Clin Nutr. 2007 Oct;86(4):1152-9. doi: 10.1093/ajcn/86.4.1152. PMID 17921396
- [Derived] Fisker AB, Lisse IM, Aaby P, Erhardt JG, Rodrigues A, Bibby BM, Benn CS. Effect of vitamin A supplementation with BCG vaccine at birth on vitamin A status at 6 wk and 4 mo of age. Am J Clin Nutr. 2007 Oct;86(4):1032-9. doi: 10.1093/ajcn/86.4.1032. PMID 17921381